CLINICAL TRIAL: NCT04589429
Title: Does Adding Nalbuphine to Intrathecal Morphine Reduce Morphine Induced Pruritus? A Randomized, Double Blind, Controlled Study.
Brief Title: Adding Nalbuphine for Control of Intrathecal Morphine Pruritus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sohair Adeeb, Principle investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 678-9/2020
Record Dates: First submitted 2020-09-27; First posted 2020-10-19 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pruritus; Pain, Postoperative; Nausea, Postoperative; Vomiting, Postoperative
Keywords: pruritus; intrathecal morphine; intrathecal nalbuphine
MeSH Terms: conditions — Pruritus; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Morphine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MN group (Active Comparator): intrathecal morphine 300 micrograms+2mg nalbuphine
  Interventions: Drug: Morphine 10 MG/ML; Drug: Nalbuphine Hydrochloride 10 MG/ML
- M group (Placebo Comparator): intrathecal morphine 300 micrograms
  Interventions: Drug: Morphine 10 MG/ML

INTERVENTIONS:
Drug: Morphine 10 MG/ML — intrathecal morphine 300 micrograms
  Other Names: morphine
Drug: Nalbuphine Hydrochloride 10 MG/ML — intrathecal nalbuphine 2mg.
  Other Names: nalbuphine
  Arms: MN group

SUMMARY:
Intrathecal morphine causes intense itching which is very bothersome. Nalbuphine antagonizes this effect when given intravenously. This trial is to find out if nalbuphine added to intrathecal morphine has an effect on morphine related pruritus while still maintaining adequate analgesia.

DETAILED DESCRIPTION:
The study will be performed in MiniaUniversity Hospitals, after obtaining approval from the local ethics committee. All patients will have a peripheral IV cannula 18 G inserted; standard non-invasive monitors will be applied. Patients undergoing major abdominal surgery will be divided into 2 groups to receive intrathecal morphine 300 micrograms with or without nalbuphine 1mg prior to anesthesia. General anesthesia is then given to patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients.
* Age 18-80yrs.
* Elective major abdominal surgery under general anesthesia.

Exclusion Criteria:

* Refusal to participate.
* Skin or systemic disease with itching. Any condition which precludes performing spinal injection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
pruritus | 2 hours postoperatively
  Pruritus score (1: no pruritus; 2: mild pruritus, treatment not requested; 3: moderate pruritus, treatment requested; 4: severe pruritus).
pruritus | 4 hours postoperatively
  Pruritus score (1: no pruritus; 2: mild pruritus, treatment not requested; 3: moderate pruritus, treatment requested; 4: severe pruritus).
pruritus | 24 hours postoperatively
  Pruritus score (1: no pruritus; 2: mild pruritus, treatment not requested; 3: moderate pruritus, treatment requested; 4: severe pruritus).

SECONDARY OUTCOMES:
postoperative pain | 2 hours postoperative
  assessed with a verbal numeric pain score(NRS) where 0: no pain; 10: worst imaginable pain
postoperative pain | 4 hours postoperative
  assessed with a verbal numeric pain score(NRS) where 0: no pain; 10: worst imaginable pain
postoperative pain | 24 hours postoperative
  assessed with a verbal numeric pain score(NRS) where 0: no pain; 10: worst imaginable pain
postoperative nausea and vomiting | 2 hours postoperative
  four-point rating score (1: no nausea or vomiting, 2: queasy, 3: severe nausea, 4: vomiting
postoperative nausea and vomiting | 4 hours postoperative
  four-point rating score (1: no nausea or vomiting, 2: queasy, 3: severe nausea, 4: vomiting
postoperative nausea and vomiting | 24 hours postoperative
  four-point rating score (1: no nausea or vomiting, 2: queasy, 3: severe nausea, 4: vomiting
Sedation | 2 hours postoperative
  four-point sedation score (1: fully awake; 2: somnolent, responds to call; 3: somnolent, responds to tactile stimulation; 4: asleep, responds to painful stimulation).
Sedation | 4 hours postoperative
  four-point sedation score (1: fully awake; 2: somnolent, responds to call; 3: somnolent, responds to tactile stimulation; 4: asleep, responds to painful stimulation).
Sedation | 24 hours postoperative
  four-point sedation score (1: fully awake; 2: somnolent, responds to call; 3: somnolent, responds to tactile stimulation; 4: asleep, responds to painful stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Sohair A Megalla, MD, Principal Investigator — Anesthesia and ICU department, Faculty of Medicine, Minia University
Locations (1):
- anesthesia&ICU department, Minya, Egypt